CLINICAL TRIAL: NCT06954428
Title: NT-301-101: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of Nasal NT-301 in Healthy Volunteers
Brief Title: Clinical Trial of Intranasal Delivery of NT-301
Acronym: APPROVE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nano PharmaSolutions Australia (Industry)
Collaborators: CMAX Clinical Research Pty Limited (Unknown); Beyond Drug Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: NT-301-101
Record Dates: First submitted 2025-03-07; First posted 2025-05-01 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Tolerability of NT-301 Nasal Spray; Pharmacokinetics of NT-301 Nasal Spray; Safety of NT-301 Nasal Spray; Performance of NT-301 Nasal Spray Device
Keywords: Safety, NT-301, tolerability, pharmacokinetics, performance of device

STUDY DESIGN:
Intervention Model Description: Single ascending dose trial in the first part (4 cohorts)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinded CRO project manager and medical affairs professional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (8):
- Placebo 1 mg (Placebo Comparator): Matching Placebo for 1 mg NT-301
  Interventions: Combination Product: NT-301 1 mg; Combination Product: Placebo 1 mg
- Placebo 2 mg (Placebo Comparator): Matching placebo for NT-301 2 mg strength
  Interventions: Combination Product: NT-301 2 mg; Combination Product: Placebo 2 mg
- NT-301 1 mg (Experimental): NT-301 nasal spray 1 mg strength
  Interventions: Combination Product: NT-301 1 mg
- NT-301 2 mg (Experimental): NT-301 nasal spray 2 mg strength
  Interventions: Combination Product: NT-301 2 mg
- Placebo 3 mg (Placebo Comparator): Matching placebo for NT-301 3 mg
  Interventions: Combination Product: Placebo 3 mg
- placebo 4 mg (Placebo Comparator): Matching placebo for NT-301 4 mg
  Interventions: Combination Product: Placebo 4 mg
- NT-301 3 mg (Active Comparator): Apomorphine nasal spray 3 mg
  Interventions: Combination Product: NT-301 3 mg
- NT-301 4 mg (Experimental): apomorphine nasal spray 4 mg
  Interventions: Combination Product: NT-301 4 mg

INTERVENTIONS:
Combination Product: NT-301 1 mg — unidose of 1 mg apomorphine through nasal spray
  Arms: NT-301 1 mg; Placebo 1 mg
Combination Product: NT-301 2 mg — unidose of 2 mg apomorphine through nasal spray
  Arms: NT-301 2 mg; Placebo 2 mg
Combination Product: Placebo 1 mg — Matching Placebo to NT-301 1 mg
  Arms: Placebo 1 mg
Combination Product: Placebo 2 mg — Matching Placebo to NT-301 2 mg
  Arms: Placebo 2 mg
Combination Product: Placebo 3 mg — Matching Placebo to NT-301 3 mg
  Arms: Placebo 3 mg
Combination Product: NT-301 3 mg — unidose apomorphine nasal spray 3 mg
  Arms: NT-301 3 mg
Combination Product: NT-301 4 mg — unidose apomorphine nasal spray 4 mg
  Arms: NT-301 4 mg
Combination Product: Placebo 4 mg — Matching placebo to NT-301 4 mg
  Arms: placebo 4 mg

SUMMARY:
The purpose of this research project is to investigate the safety and tolerability of an approved drug (Apomorphine) when administered as a nasal powder spray formulation (NT-301) as well as collect information on how NT-301 moves into, through and out of your body, called Pharmacokinetics.

DETAILED DESCRIPTION:
Single Ascending Dose (SAD)- 4 groups will receive a single dose only. Each group receiving a dose higher than the previous cohort. Some participants will get a nasal spray containing NT-301 and others will get a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged between 18 and 60 years of age, inclusive at the time of signing the informed consent document.
2. Body weight ≥50 kg and body mass index (BMI) within the range of 18 to 32 kg/m2 inclusive at screening.
3. Woman of childbearing potential (WOCBP) or fertile male participants must agree to use an acceptable method of contraception from the start of Screening until 90 days (male participants) or 60 days (female participants) after the final study visit.
4. WOCBP must have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to administration of the first dose of study intervention (including domperidone) and be willing to have additional pregnancy tests, as required, throughout the study.
5. Participants must be in good general health, as demonstrated at screening and prior to first administration of any study intervention (including domperidone) by the absence of clinically significant (in the opinion of the Investigator) abnormalities based on a medical evaluation including review of medical history, physical examination, safety laboratory tests, vital signs, 12-lead ECG monitoring.

   Note: It is the responsibility of the Investigator to assess the clinical significance of any abnormality/ies; however, consultation with the MM may be warranted.
6. Normal vital signs after ≥5 min resting in supine position:

   1. ≥90 mmHg and ≤160 mmHg systolic blood pressure (SBP)
   2. ≥50 mmHg and ≤95 mmHg diastolic blood pressure (DBP)
   3. ≥ 45 bpm and ≤100 bpm heart rate (HR)
   4. Body temperature (tympanic) ≥35.5°C and ≤37.7°C
7. No clinically significant changes and/or associated symptoms considered related to orthostatic hypotension when measuring blood pressure (BP) and pulse rate (PR) within 2 min of standing from a supine position.
8. Triplicate 12-lead ECG, taken after ≥5 min in a supine, position, with a QT interval corrected using the Fridericia method (QTcF) ≤ 450 msec for males and ≤ 470 msec for females, PR interval ≤ 220 msec or QRS duration ≤ 120 msec or history of long QT syndrome and no clinically significant abnormalities as judged by the Investigator (or qualified designee).
9. Willing and able to be confined at the CRU for the study period and adhere to overall study visit schedule, procedures and other protocol requirements, as assessed by the Investigator (or qualified designee).
10. Understands and voluntarily signs an informed consent document prior to any study related assessments/procedures being conducted.

Exclusion Criteria:

1. Any significant medical condition, physical or psychiatric illness or history of depression that could, in the Investigator's (or qualified designee) opinion, compromise the participant's safety or interfere with the completion of this study.
2. History of clinically significant CNS, cardiac, pulmonary, metabolic, renal, hepatic, or gastrointestinal (GI) conditions including gastric bypass or other weight loss surgical procedure.
3. Any condition including the presence of laboratory abnormalities, which according to the Investigator (or qualified designee), places the participant at unacceptable risk if they were to participate in the study or may confound the ability to interpret data from the study. This includes the presence of uncontrolled current illness (e.g., an infection), a viral infection, seasonal allergy, or concurrent skin rash.
4. Any nasal condition, including nasal congestion, physical blockage of either nostril, deviated septum, structural or anatomical nasal conditions or nasal surgery in the last 6 months. Use of topical nasal medications (e.g., acute or chronic use of prescription or over the counter nasal sprays) that may affect the administration or absorption of the study drug.
5. Use of 5HT3 antagonists, drugs known to prolong QTc, and use of antihypertensives.
6. The participant has a medical history of or a positive blood test for human immunodeficiency virus (HIV: HIV, anti-HIV1 and anti-HIV2 antibodies), hepatitis C virus (HCV, anti-HCV antibodies), or hepatitis B surface antigen (HBsAg) at screening.
7. Aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT), serum creatine, or total bilirubin >1.5x the upper limit of normal (ULN). These laboratory tests may be repeated once if they are abnormal on first screening, and if there is a medical reason to believe the results may be inaccurate. If the repeat test is within the normal range, the participant may be included in the study only if the Investigator (or qualified designee) considers that the previous finding will not compromise the participant's safety and will not interfere with the interpretation of safety data.
8. A positive drug or alcohol screen. A positive drug or alcohol screen test result may be verified by re-testing at the discretion of the Investigator (or qualified designee), with up to 1 false positive result permitted.
9. History of regular alcohol consumption within 6 months of screening defined as an average weekly intake of >21 units. One unit is equivalent to 10 g of alcohol and the following can be used as a guide: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (30 mL) measure of spirits.
10. The participant is unwilling to abstain from alcohol consumption from 24 h prior to treatment with any study intervention (including domperidone) and until discharge from the CRU, and for 24 h prior to all other outpatient visits to the CRU.
11. The participant is pregnant or planning to become pregnant within 90 days of the study or is breastfeeding.
12. Major surgery within 4 weeks of screening that could interfere with, or for which the treatment might interfere with, the conduct of the study, or that would pose an unacceptable risk to the participant in the opinion of the Investigator (or qualified designee).
13. Use of tobacco or nicotine products exceeding 5 cigarettes (or equivalent) per week in any form within 30 days prior to treatment with any study intervention (including domperidone), or unwillingness to refrain from smoking, vaping, or using any nicotine products for at least 48 h prior to dosing with any study intervention (including domperidone), the confinement period, and any follow up visits.
14. The participant uses or is planning to use any prescription or non-prescription medications (with the exception of hormonal contraceptives), herbal and dietary supplements, within 5 days or 5 half-lives (whichever is longer) prior to treatment with any study intervention (including domperidone), unless in the opinion of the PI, local MM and Sponsor medical representative, the medication is not expected to interfere with the study procedures or compromise participant safety
15. Participation in a clinical trial and receipt of an investigational medication within 90 days, 5 half-lives (if known) or twice the duration of the biological effect of any medication, whichever is longer, prior to the first dose of study intervention.
16. Use of any strong CYP450-3A4/5 inhibiting or inducing agents within 14 days of dosing with any study intervention (including domperidone) and for the duration of the study.
17. Consumption of grapefruit, grapefruit juice, star fruit, oranges, orange juice, Seville oranges, within 14 days prior to dosing with any study intervention (including domperidone) and participant is unwilling to abstain from consumption of these products until after discharge from the CRU.
18. Participant is unwilling to abstain from the consumption of caffeine and/or xanthine containing products (e.g., coffee, tea, chocolate, and caffeine containing sodas, etc.) from time of admission to the CRU on Day -1 until after discharge from the CRU.
19. Known sensitivity to any study intervention, including NT-301, apomorphine HCl and domperidone.
20. Loss or donation of whole blood (>499 mL) within 3 months and/or plasma donation within 2 weeks, prior to dosing with any study intervention (including domperidone), or intention to donate blood or blood products during the study.
21. The participant has a history of cancer, with the exception of basal cell carcinoma or in situ cervical cancer that has been in remission for ≥5 years prior to first dose of study treatment.
22. Participants with a pre-disposition to nausea and vomiting (e.g., history of severe travel sickness).
23. The participant is unwilling or unable to follow protocol requirements, including domperidone self-administration and diary completion, and attendance at follow up visit(s), or otherwise unsuitable for study participation in the opinion of the Investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
Safety of NT-301 | Enrollment to 7 days after dosing
  Laboratory safety data
Tolerability of NT-301 | Enrollment to 7 day post dose
  Nasal examinations by the Quantitative Scoring Scale - Nasal Mucosa (QSS-NM): range 0 to 34.

SECONDARY OUTCOMES:
Pharmacokinetics of Apomorphine | Predosing to 24 hours post dosing
  Cmax (ng/mL)
Pharmacokinetics of Apomorphine | Predose to 24 hour post dose
  Area under curve (AUC): ng*hr/mL
Pharmacokinetics of Apomorphine | Predose to 24 hour post dose
  Tmax: in hour

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - CMAX Clinical Research Center Pty Limited, Adelaide, South Australia
  - CMAX, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: Undecided